CLINICAL TRIAL: NCT05919758
Title: The Value of Complementary Right-sided Hemicolectomy for Pediatric Patients With High-risk Neuroendocrine Tumors (NETs) of the Appendix; Towards the Development of an (Inter-) National Consensus Guideline for the Pediatric Population.
Brief Title: Value of Right-sided Hemicolectomy for Chldren With High-risk Neuroendocrine Tumors of the Appendix
Acronym: NETkids
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Ramon Gorter, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_169#21.184
Record Dates: First submitted 2023-05-08; First posted 2023-06-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Neoplasms; Appendix Cancer
MeSH Terms: conditions — Neoplasms; Appendiceal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate the beneficial value of complementary surgery for appendiceal neuro-endocrine tumours in children.

.

DETAILED DESCRIPTION:
Aim Current guidelines recommend complementary right-sided hemicolectomy for high-risk (pT2(with risk factors)/pT3) neuro-endocrine tumors (NET) of the appendix (based on adult studies). In contrast to adults, high-risk NET of the appendix in children seems to be a relatively benign disease with high disease-free survival (100% versus 70-80% in adults), but high quality data are lacking. Therefore these recommendations are now being questioned. We aim to investigate the value of complementary right-sided hemicolectomy for children with high-risk NET of the appendix. Ultimately leading to the development of a consensus guideline and solid information for patients/parents.

Plan of investigation In order to generate big data, an international historical cohort study is planned to compare complementary right-sided hemicolectomy with appendectomy alone for children with high-risk NET of the appendix. Results will be CONFIDENTIAL used by an international expert group to formulate treatment recommendations. Subsequently, these recommendations will be tested in an international Delphi study in order to develop a consensus guideline on the treatment of pediatric high-risk NET of the appendix.

Expected results The cohort study will generate high quality information on overall/disease-free survival, recurrence, complications, costs, and hr-QoL. Recommendations made will be tested in a Delphi study; not only on the beneficial value of complementary right-sided hemicolectomy, but also on follow-up protocols and preoperative work-up. Ultimately, an international consensus guideline that redefines low-risk and high-risk NET of the appendix will be developed, leading to global de-escalation and uniformity of treatment.

Relevance for childhood cancer Results are relevant for pediatric oncologists/surgeons/gastro-enterologists across the world, as redefining low-risk and high-risk patient groups, will lead to de-escalation of treatment. Furthermore, QoL of child and parents can be improved by reducing exposure to complications after complementary right-sided hemicolectomy, and by reducing the fear of recurrence by obtaining high-quality data to accurately inform patients and parents.

ELIGIBILITY:
Inclusion Criteria:

* All patients that were treated for an appendiceal NET before the age of 18 years old
* Time period: 1990-2020

Exclusion Criteria:

* Other appendiceal malignancies/tumours, for example:
* goblet cell carcinoma
* adenocarcinoma
* neuroendocrine carcinoma

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: All patients treated for an appendiceal neuro endocrine tumour before the age of 18 during 1990 and 2020
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Disease free survival rate | cross-sectional design. follow-up will be done in 2023/2024
  defined as alive and free of recurrence of NET at telephone follow-up performed for this study purpose
Recurrence rate | cross-sectional design. follow-up will be done in 2023/2024
  defined as histopathologically proven metastasis/residual tumor at appendiceal stump of NET after a disease free period

SECONDARY OUTCOMES:
Overall survival rate | cross-sectional design. follow-up will be done in 2023/2024
  defined as alive at telephone follow-up performed for this study purpose
Complications directly related to primary and secondary treatment divided into major and minor complications according to Clavien-dindo. | cross-sectional design. follow-up will be done in 2023/2024
  Complications include, but are not limited to:
  * Intra-abdominal abscess, defined as a radiologically confirmed accumulation of purulent fluid in a walled-off space within the abdominal cavity.
  * (Adhesive) bowel obstruction requiring readmission (diagnosis based on clinical signs and symptoms such as a history of constipation, nausea, vomiting and distended abdomen)
  * Superficial Surgical Site Infection, as defined by the CDC criteria. (see table 1.)
  * Deep Surgical Site Infection, as defined by the CDC criteria.
Number of hospital readmission for complications related to treatment of NET | cross-sectional design. follow-up will be done in 2023/2024
  see title
Length of hospital stay | cross-sectional design. follow-up will be done in 2023/2024
  initial and total length of stay
number of imaging studies performed for follow-up of NET | cross-sectional design. follow-up will be done in 2023/2024
  ultrasound, computed tomography (CT), magnetic resonance imaging (MRI), octreotide scintigraphy, PET-CT
Number of outpatient check-ups(regular visits / telephone call) for follow-up of NET | cross-sectional design. follow-up will be done in 2023/2024
  see title
Health related Quality of Life at follow-up moment for this study | cross-sectional design. follow-up will be done in 2023/2024
  measured by the PedsQL(generic)
Health related Quality of Life at follow-up moment for this study | cross-sectional design. follow-up will be done in 2023/2024
  measured by the QLQ-C30(generic)
Health related Quality of Life at follow-up moment for this study | cross-sectional design. follow-up will be done in 2023/2024
  measured by the QLQ-GINET-21 questionnaire(disease specific)

CONTACTS AND LOCATIONS:
Overall Officials: Ramon R Gorter, MD PhD, Study Chair — Amsterdam UMC, department of pediatric surgery
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, Netherlands

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared with other researchers. Collaborating institution will however enter participant data in a coded/pseudonimyzed manner in Castor EDC database.